CLINICAL TRIAL: NCT01075971
Title: Evaluation of Preference Between Two Buprenorphine Sublingual Formulations, After a Switch From the Marketed Tablet (Subutex®) to the New Fast Dissolving Tablet (FDT), in Opioid-dependent Patients With Buprenorphine Maintenance Therapy
Brief Title: Study of Two Formulations of Buprenorphine HCl in Opioid-dependent Subjects on Buprenorphine Maintenance Therapy (Study P04451) (COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Collaborators: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04451
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Opioid Dependency
Keywords: Buprenorphine tablet; Fast dissolving tablet; Opioid dependant patients
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine hydrochloride (Experimental)
  Interventions: Drug: Buprenorphine hydrochloride marketed sublingual tablet (Subutex); Drug: Buprenorphine hydrochloride fast dissolving tablet (FDT)

INTERVENTIONS:
Drug: Buprenorphine hydrochloride marketed sublingual tablet (Subutex) — 8 mg or 16 mg daily, sublingual route on Days 1 and 2
  Other Names: Subutex®
Drug: Buprenorphine hydrochloride fast dissolving tablet (FDT) — 8 mg or 16 mg daily, sublingual route on Days 3, 4, and 5

SUMMARY:
This is a multi-center, open-label, preference study of two sublingual formulations of buprenorphine HCl, in opioid-dependent patients on buprenorphine maintenance therapy.

The objectives of this study are to evaluate the overall preference between two buprenorphine sublingual formulations, after a switch from the marketed tablet (Subutex®) to the new fast dissolving tablet (FDT), in opioid-dependent patients with buprenorphine 8 mg or 16 mg daily maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Patients must be at least (≥) 18 years of age, of either sex.
* Patients treated for opioid dependence with Subutex®, with a stable dosage of 8 mg or 16 mg daily, and respecting the legal drug attachments.
* Patients must understand and be able to adhere to the dosing and visit schedules, and agree to report concomitant medications / products and adverse events to the investigator or designee.
* Women of childbearing potential (includes women who are less than one year postmenopausal and women who become sexually active) must be using or agree to use an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterile (e.g., hysterectomy or tubal ligation).
* Women of childbearing potential should be counseled in the appropriate use of birth control while in this study. Women who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.
* Women of childbearing potential must have a urine pregnancy test with negative result within 2 weeks prior to inclusion (as performed under control of the investigator or designee).

Exclusion Criteria:

* Patients refusing to take the daily dose of the study medication under control in the center.
* Patients unable to complete the evaluations.
* Women who are pregnant or nursing.
* Patients with a history of hypersensitivity to buprenorphine hydrochloride or any excipient of one of its formulations.
* Patients with a current evidence of alcohol abuse.
* Patients with severe respiratory dysfunction, severe hepatic dysfunction, acute alcohol intoxication or delirium tremens.
* Initiation or increase in the dose, within the past 7 days or scheduled during the study, of a treatment with:

  * benzodiazepines,
  * other depressants of the central nervous system: other morphine derivatives (analgesics, antitussives), certain antidepressive agents, sedative H1 antihistamines, barbiturates, benzodiazepines, anxiolytics other than benzodiazepines, neuroleptics, clonidine and clonidine-like agents,
  * monoamine oxydase [MAO] inhibitors.
* Patients who have any current evidence of clinically significant hematopoietic, metabolic, cardiovascular, immunologic, neurologic, hematological, gastrointestinal, hepatic, renal, psychiatric, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the investigator, may interfere with the study evaluations or affect patient safety.
* Patients who have used any investigational product within 30 days prior to enrollment.
* Patients participating in another trial at the same time.
* Patients intending to donate blood during the study or within 3 months after study completion.
* Patients in the exclusion period of the "Fichier National des personnes qui se prêtent à des recherches biomédicales sans bénéfice individuel direct" (National Index of persons participating in biomedical researches without direct individual benefit, or National Index of volunteers).
* Patients without Social Security number, or whose maximum annual compensation (3,800 €) has been exceeded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine Hydrochloride: 8 or 16 mg daily for 5 days; marketed sublingual tablet on Days 1 and 2, fast dissolving tablet (FDT) on Days 3, 4, and 5
Period: Overall Study
Arm/Group | Buprenorphine Hydrochloride
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine Hydrochloride
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.94 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 42
Region of Enrollment [Number; unit: participants]
  France | 52

OUTCOME MEASURES:

1. Primary Outcome: The Overall Preference Between Two Buprenorphine Sublingual Formulations, After a Switch From the Marketed Tablet (Subutex®) to the New Fast Dissolving Tablet (FDT), in Opioid-dependent Patients With Buprenorphine 8 mg or 16 mg Daily Maintenance Therapy.
Description: Patient's overall satisfaction on Day 1 to Day 5 postdose. Marketed sublingual tablet (Marketed SL): Days 1 and 2; Fast dissolving tablet (FTD): Days 3, 4, and 5. Within 1 hour after complete dissolution of the tablet(s), overall satisfaction towards the study treatment was to be scored by the patient himself / herself using a 10-cm visual analogic scale (VAS) ranging from "Not at all satisfied" (score = 0) to "Totally satisfied" (score = 10).
Time Frame: Daily, Day 1 to Day 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Buprenorphine Hydrochloride
Number analyzed (Participants) | 52
Score on a scale
  Day 1 Marketed SL | 6.01 (2.42)
  Day 2 Marketed SL | 5.91 (2.24)
  Day 3 FTD | 7.73 (1.77)
  Day 4 FTD | 7.75 (1.74)
  Day 5 FTD | 7.72 (1.76)
  Overall SL formulation | 5.96 (2.32)
  Overall FTD formulation | 7.73 (1.74)
Statistical Analysis 1: Comparison: Buprenorphine Hydrochloride; Test type: Superiority or Other; p < 0.0001, Analysis of variance — Analysis of variance with repeated measurements (daily scores from day 1 to day 5) for the whole set of patients was performed adjusted on the formulation (SL vs. FDT). Other independent factors were the subject and the day; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [1.35 to 2.19]

ADVERSE EVENTS:
Time Frame: All adverse events, including AEs that started before the first dose.
Arm/Group | Buprenorphine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 3/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Hydrochloride (N=52)
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's representative will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.